CLINICAL TRIAL: NCT07329270
Title: Postpartum Depression Prevention Program in Disaster-Affected Regions
Brief Title: A Trauma-Informed Primary Health Care Intervention to Prevent Postpartum Depression After Disaster
Acronym: TIPPDP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, Zeynep Şimşek, Professor of Public Health and Social Work / Dean, Faculty of Health Sciences, Istanbul Bilgi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BAP-2023.02.002; TUBİTAK424K188 (Other Grant/Funding Number: Scientific Research Projects Unit (BAP) of İstanbul Bilgi University and Scientific and Technological Research Council)
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Postpartum Depression (PPD)
Keywords: postpartum depression | trauma-informed care | disaster response | maternal mental health | primary health care | resilience | Türkiye earthquakes
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: Participants were assigned in parallel to either a trauma-informed postpartum depression prevention program or to usual postpartum care. The intervention was developed using findings from an initial qualitative phase and evaluated using an experimental design.
Who Masked: Participant
Masking Description: Participants were masked to group assignment. Due to the nature of the psychosocial intervention, care providers were not masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trauma-Informed Postpartum Depression Prevention Program (Experimental): Participants in this arm received a trauma-informed postpartum depression prevention program developed by the research team. The program was informed by findings from an initial qualitative phase using interpretative phenomenological analysis and was integrated into routine primary health care services in earthquake-affected regions. The intervention focused on early identification of psychological distress, psychoeducation, emotional support, strengthening coping skills, and enhancing social support.
  Interventions: Behavioral: Trauma-Informed Preventive Intervention
- No Intervention / Usual Care (No Intervention): Participants in this arm received usual postpartum care provided through routine primary health care services without a structured trauma-informed mental health prevention component.

INTERVENTIONS:
Behavioral: Trauma-Informed Preventive Intervention — This is a newly developed trauma-informed postpartum depression prevention program designed for women living in earthquake-affected regions. The program was developed by the research team based on qualitative findings from in-depth interviews with postpartum women analyzed using interpretative phenomenological analysis. It was delivered within primary health care settings by trained health care professionals and included psychoeducation, emotional support, coping skills enhancement, and facilitation of social support and referral when needed.
  Arms: Trauma-Informed Postpartum Depression Prevention Program

SUMMARY:
Postpartum depression is a common mental health problem that can affect women after childbirth and may have long-lasting consequences for both mothers and infants. The risk of postpartum depression is substantially higher in disaster-affected regions due to exposure to trauma, loss, displacement, disruption of health services, and ongoing psychosocial stressors.

This study aimed to develop and evaluate a trauma-informed postpartum depression prevention program for women living in earthquake-affected regions of Türkiye using a sequential mixed-methods design. In the first phase, the program was developed based on qualitative findings obtained through in-depth interviews with postpartum women. In the second phase, the effectiveness of the newly developed program was tested using an experimental design.

During the qualitative phase, in-depth interviews were conducted with 24 postpartum women, and data were analyzed using interpretative phenomenological analysis (IPA) to explore women's lived experiences, perceived needs, and priorities related to mental health and psychosocial support after childbirth in a disaster context. The findings from this phase informed the content, structure, and delivery of the trauma-informed prevention program.

In the quantitative phase, the program was evaluated through a randomized controlled trial. Eligible postpartum women were randomly assigned either to the trauma-informed prevention program or to a comparison group receiving usual primary health care services. Postpartum depressive symptoms were assessed using validated measures.

The primary objective of the study was to evaluate the effectiveness of the trauma-informed program in reducing postpartum depressive symptoms. The findings are expected to contribute to evidence-based, trauma-informed approaches for preventing postpartum depression in disaster-affected settings.

DETAILED DESCRIPTION:
Women living in disaster-affected regions face increased vulnerability to postpartum depression due to exposure to traumatic events, loss of social and material resources, disruptions in health care delivery, and prolonged uncertainty. Addressing postpartum mental health in such contexts requires interventions that are both evidence-based and responsive to women's lived experiences.

This study employed a sequential mixed-methods design to develop and evaluate a trauma-informed postpartum depression prevention program for women living in earthquake-affected regions of Türkiye. The study consisted of two consecutive phases: a qualitative program development phase and a quantitative experimental evaluation phase.

In the first phase, the trauma-informed postpartum depression prevention program was developed by the research team based on qualitative data collected from 24 postpartum women. In-depth, semi-structured interviews were conducted to explore participants' lived experiences of the postpartum period in a disaster context, perceived psychosocial needs, sources of distress and support, and expectations from health care services. The qualitative data were analyzed using interpretative phenomenological analysis (IPA), allowing for an in-depth understanding of participants' subjective experiences and meaning-making processes. The findings from this phase directly informed the content, focus, and delivery strategies of the intervention.

In the second phase, the effectiveness of the newly developed program was evaluated using an experimental design. Eligible postpartum women were recruited through primary health care services and randomly assigned to either the intervention group, which received the trauma-informed postpartum depression prevention program, or a comparison group receiving usual postpartum care. The intervention was delivered within routine primary health care settings by trained health care professionals.

The primary outcome of the study was postpartum depressive symptoms, assessed using validated screening instruments at predefined follow-up points. Secondary outcomes included measures of perceived social support, stress and coping perception. Data collection and outcome assessments were conducted in accordance with the study protocol.

By combining qualitative insights from postpartum women with rigorous experimental testing, this study aimed to generate robust evidence on the development and effectiveness of trauma-informed preventive interventions for postpartum depression in disaster-affected settings. The findings are intended to inform maternal mental health practice, program development, and public health policy in disaster and post-disaster contexts.

ELIGIBILITY:
Inclusion Criteria:

Postpartum women aged 18 years or older

Having an infant younger than 60 days at the time of enrollment

Living in earthquake-affected regions of Türkiye

Receiving routine postpartum follow-up through primary health care services

Able to communicate in Turkish

Provided written informed consent

Exclusion Criteria:

History of a diagnosed psychiatric disorder prior to the current postpartum period

Severe medical conditions requiring specialized care

Cognitive impairment or any con

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Postpartum Depressive Symptoms | Baseline and at infant age 6 months.
  Postpartum depressive symptoms were assessed using the Edinburgh Postnatal Depression Scale (EPDS), a validated 10-item self-report instrument widely used for screening depressive symptoms during the postpartum period. Higher scores indicate greater severity of depressive symptoms. The primary outcome was the change in EPDS scores from baseline to six months post-intervention.

SECONDARY OUTCOMES:
Perceived Stress | Baseline and at infant age 6 months.
  Perceived stress was assessed using a self-report item asking participants how often they felt stressed during the past week, rated on a five-point scale ranging from "never" to "very often." Higher scores indicate higher perceived stress levels.

OTHER OUTCOMES:
Coping Perception | Baseline and at infant age 6 months.
  Coping perception was assessed using a self-report item evaluating how often participants felt unable to cope with their problems during the past week, rated on a five-point Likert-type scale. Higher scores reflect stronger perceived coping ability.
Perceived social support | Baseline and at infant age 6 months.
  Perceived social support was assessed using the Multidimensional Scale of Perceived Social Support (MSPSS), which measures perceived support from family, friends, and a significant other. Higher scores indicate greater perceived social support.

CONTACTS AND LOCATIONS:
Locations (1):
- Narlıca 2 No'lu Family Physician Center, Hatay, Antakya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The dataset includes sensitive mental health information collected from postpartum women living in disaster-affected regions, and data sharing is restricted due to ethical and confidentiality considerations.

REFERENCES:
- [Background] Manuscript under peer review.